CLINICAL TRIAL: NCT07033611
Title: Effects of Creatine Supplementation in Sarcopenic and Non-sarcopenic Patients on Chronic Hemodialysis
Brief Title: Effects of Short Term Creatine Supplementation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carla Basualto Alarcón (Other)
Responsible Party: Sponsor-Investigator, Carla Basualto Alarcón, Associate Professor, U Aysen. MD., MSc., PhD., Universidad de Aysén
Organization: Universidad de Aysén (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORD252023
Record Dates: First submitted 2025-06-02; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dialysis; Complications; Performance Enhancing Product Use
Keywords: dialysis; poor physical performance; creatine; body composition; Short Physical Performance Battery (SPPB); handgrip test
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Functional assessments and bioelectrical impedance analysis conducted pre- and post-creatine supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre creatine and post (Experimental): patients before and after creatine suplemmentation
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: Creatine — Five grams of creatine were administered to each patient daily for eight weeks.

SUMMARY:
Adult patients undergoing chronic dialysis therapy for at least three months were selected. A physical function assessment was conducted, including the Short Physical Performance Battery (SPPB) and a handgrip strength test. Additionally, a bioelectrical impedance analysis was performed. Subsequently, 5 grams of creatine were administered daily for a period of eight weeks, after which the same assessments were repeated. The results were then analyzed to identify any differences in the tests, aiming to detect potential changes following creatine supplementation.

DETAILED DESCRIPTION:
Adult patients undergoing chronic dialysis therapy for at least three months were selected, primarily based on their good adherence to pharmacological and dialysis treatment regimens. A physical function assessment was conducted, including the Short Physical Performance Battery (SPPB) and a handgrip strength test. Additionally, a bioelectrical impedance analysis was performed.

All participants were informed that creatine would be administered and provided written informed consent. The study protocol was approved by the local ethics committee.

Creatine supplementation consisted of 5 grams per day for eight weeks. On dialysis days, the dose was administered immediately after the dialysis session. On non-dialysis days, patients were responsible for self-administering the creatine at home. The creatine was diluted in 100 mL of water before ingestion.

All assessments were conducted the day following the second dialysis session of the week-on Thursday or Friday, depending on the patient's schedule. There was no control group so pre-creatine measurements were considered as the basal (control) state. Measurements were taken before and after the creatine supplementation period in the same patients. The data were analyzed to evaluate changes in the outcomes following creatine use.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to provide informed consent
* At least three months on chronic dialysis therapy
* No physical impairments that would prevent completion of the SPPB or bioelectrical impedance analysis

Exclusion Criteria:

* Pregnancy
* Use of any nutritional supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Compare Short Physical Performance Battery (SPPB) before and after 8 weeks of creatine use | eigth weeks
  To compare the physical functionality status of selected patients, as assessed by the Short Physical Performance Battery (SPPB), before and after eight weeks of creatine supplementation. Scale range between 0-12 points. Higher points mean a better outcome (higher physical functionality).

SECONDARY OUTCOMES:
Compare hand grip strength as assessed by a hand dynamometer, before and after eight weeks of creatine supplementation | eigth weeks
  compare changes in muscle strength, measured using a hand dynamometer.
Compare body composition: skeletal muscle mass, estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in skeletal muscle mass (Kg), estimated by bioimpedance analysis before and after eight weeks of creatine supplementation
Compare body composition: fat free mass, estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in fat free mass (Kg), estimated by bioimpedance analysis before and after
Compare body composition: total body water (Lt), estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in tota body water (Lt), estimated by bioimpedance analysis before and after
Compare body composition: extracellular water (Lt), estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in extracellular water (Lt), estimated by bioimpedance analysis before and after
Compare body composition: intracellular water (Lt), estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in intracellular water (Lt), estimated by bioimpedance analysis before and after
Compare body composition: phase angle (degrees), estimated by bioimpedance analysis before and after eight weeks of creatine supplementation | eigth weeks
  Compare changes in phase angle (degrees), estimated by bioimpedance analysis before and after

CONTACTS AND LOCATIONS:
Overall Officials: Carla Basualto-Alarcón, PhD, Principal Investigator — Universidad de Aysén
Locations (1):
- Hospital de Puerto Aysen, Puerto Aisén, Región de Aysen, Chile

IPD SHARING:
Plan to Share IPD: Yes
At the time of paper submission, all data will be shared in an anonymized form, as supplementary material.

REFERENCES:
- [Background] Wallimann T, Riek U, Moddel M. Intradialytic creatine supplementation: A scientific rationale for improving the health and quality of life of dialysis patients. Med Hypotheses. 2017 Feb;99:1-14. doi: 10.1016/j.mehy.2016.12.002. Epub 2016 Dec 7. PMID 28110688
- [Background] Johansen KL, Chertow GM, Ng AV, Mulligan K, Carey S, Schoenfeld PY, Kent-Braun JA. Physical activity levels in patients on hemodialysis and healthy sedentary controls. Kidney Int. 2000 Jun;57(6):2564-70. doi: 10.1046/j.1523-1755.2000.00116.x. PMID 10844626
- [Background] Jain N, Bansal R, Saxena S, Sharma S, Raju SB. Predictors of functional impairment and mortality in patients on maintenance hemodialysis. Semin Dial. 2024 Mar-Apr;37(2):138-144. doi: 10.1111/sdi.13173. Epub 2023 Aug 24. PMID 37615221
- [Background] Nowicka M, Gorska M, Edyko K, Szklarek-Kubicka M, Kazanek A, Prylinska M, Niewodniczy M, Kostka T, Kurnatowska I. Association of Physical Performance, Muscle Strength and Body Composition with Self-Assessed Quality of Life in Hemodialyzed Patients: A Cross-Sectional Study. J Clin Med. 2022 Apr 20;11(9):2283. doi: 10.3390/jcm11092283. PMID 35566409
- [Background] Torino C, Manfredini F, Bolignano D, Aucella F, Baggetta R, Barilla A, Battaglia Y, Bertoli S, Bonanno G, Castellino P, Ciurlino D, Cupisti A, D'Arrigo G, De Paola L, Fabrizi F, Fatuzzo P, Fuiano G, Lombardi L, Lucisano G, Messa P, Rapana R, Rapisarda F, Rastelli S, Rocca-Rey L, Summaria C, Zuccala A, Tripepi G, Catizone L, Zoccali C, Mallamaci F; EXCITE Working Group. Physical performance and clinical outcomes in dialysis patients: a secondary analysis of the EXCITE trial. Kidney Blood Press Res. 2014;39(2-3):205-11. doi: 10.1159/000355798. Epub 2014 Jul 29. PMID 25118076
- [Background] Morishita S, Tsubaki A, Shirai N. Physical function was related to mortality in patients with chronic kidney disease and dialysis. Hemodial Int. 2017 Oct;21(4):483-489. doi: 10.1111/hdi.12564. Epub 2017 Apr 18. PMID 28418625
- [Background] Kavanagh NT, Schiller B, Saxena AB, Thomas IC, Kurella Tamura M. Prevalence and correlates of functional dependence among maintenance dialysis patients. Hemodial Int. 2015 Oct;19(4):593-600. doi: 10.1111/hdi.12286. Epub 2015 Mar 2. PMID 25731070
- [Background] Delanaye P, Quinonez K, Buckinx F, Krzesinski JM, Bruyere O. Hand grip strength measurement in haemodialysis patients: before or after the session? Clin Kidney J. 2018 Aug;11(4):555-558. doi: 10.1093/ckj/sfx139. Epub 2017 Dec 19. PMID 30090629
- [Background] Hultman E, Soderlund K, Timmons JA, Cederblad G, Greenhaff PL. Muscle creatine loading in men. J Appl Physiol (1985). 1996 Jul;81(1):232-7. doi: 10.1152/jappl.1996.81.1.232. PMID 8828669
- [Background] Kim HJ, Kim CK, Carpentier A, Poortmans JR. Studies on the safety of creatine supplementation. Amino Acids. 2011 May;40(5):1409-18. doi: 10.1007/s00726-011-0878-2. Epub 2011 Mar 12. PMID 21399917
- [Background] Liu CK, Seo J, Lee D, Wright K, Tamura MK, Moye JA, Bean JF, Weiner DE. Mobility in Older Adults Receiving Maintenance Hemodialysis: A Qualitative Study. Am J Kidney Dis. 2022 Apr;79(4):539-548.e1. doi: 10.1053/j.ajkd.2021.07.010. Epub 2021 Aug 20. PMID 34419517
- [Background] Bao Y, Dalrymple L, Chertow GM, Kaysen GA, Johansen KL. Frailty, dialysis initiation, and mortality in end-stage renal disease. Arch Intern Med. 2012 Jul 23;172(14):1071-7. doi: 10.1001/archinternmed.2012.3020. PMID 22733312
- [Background] Kang SH, Do JY, Kim JC. Impedance-derived phase angle is associated with muscle mass, strength, quality of life, and clinical outcomes in maintenance hemodialysis patients. PLoS One. 2022 Jan 12;17(1):e0261070. doi: 10.1371/journal.pone.0261070. eCollection 2022. PMID 35020730
- [Background] Kreider RB, Jager R, Purpura M. Bioavailability, Efficacy, Safety, and Regulatory Status of Creatine and Related Compounds: A Critical Review. Nutrients. 2022 Feb 28;14(5):1035. doi: 10.3390/nu14051035. PMID 35268011
- [Background] Bucar Pajek M, Cuk I, Mlinsek G, Osredkar J, Pajek J. Physical function and 25-hydroxyvitamin D in dialysis patients - lessons learned from the Slovenian DIAGIB study. Clin Nephrol. 2017 Supplement 1;88(13):48-52. doi: 10.5414/CNP88FX12. PMID 28601123
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Beberashvili I, Azar A, Sinuani I, Shapiro G, Feldman L, Stav K, Sandbank J, Averbukh Z. Bioimpedance phase angle predicts muscle function, quality of life and clinical outcome in maintenance hemodialysis patients. Eur J Clin Nutr. 2014 Jun;68(6):683-9. doi: 10.1038/ejcn.2014.67. Epub 2014 Apr 16. PMID 24736681
- [Background] Garlini LM, Alves FD, Ceretta LB, Perry IS, Souza GC, Clausell NO. Phase angle and mortality: a systematic review. Eur J Clin Nutr. 2019 Apr;73(4):495-508. doi: 10.1038/s41430-018-0159-1. Epub 2018 Apr 26. PMID 29695763
- [Background] Uchida J, Suzuki Y, Imamura K, Yoshikoshi S, Nakajima T, Fukuzaki N, Harada M, Kamiya K, Matsuzawa R, Matsunaga A. The Association of Short Physical Performance Battery With Mortality and Hospitalization in Patients Receiving Hemodialysis. J Ren Nutr. 2024 May;34(3):235-242. doi: 10.1053/j.jrn.2023.10.010. Epub 2023 Nov 3. PMID 37923149
- [Background] van der Veen Y, Post A, Kremer D, Koops CA, Marsman E, Appeldoorn TYJ, Touw DJ, Westerhuis R, Heiner-Fokkema MR, Franssen CFM, Wallimann T, Bakker SJL. Chronic Dialysis Patients Are Depleted of Creatine: Review and Rationale for Intradialytic Creatine Supplementation. Nutrients. 2021 Aug 6;13(8):2709. doi: 10.3390/nu13082709. PMID 34444869
- [Background] Post A, Schutten JC, Kremer D, van der Veen Y, Groothof D, Sotomayor CG, Koops CA, de Blaauw P, Kema IP, Westerhuis R, Wallimann T, Heiner-Fokkema MR, Bakker SJL, Franssen CFM. Creatine homeostasis and protein energy wasting in hemodialysis patients. J Transl Med. 2021 Mar 20;19(1):115. doi: 10.1186/s12967-021-02780-y. PMID 33743724
- [Background] Post A, Tsikas D, Bakker SJL. Creatine is a Conditionally Essential Nutrient in Chronic Kidney Disease: A Hypothesis and Narrative Literature Review. Nutrients. 2019 May 10;11(5):1044. doi: 10.3390/nu11051044. PMID 31083291
- [Background] Marini ACB, Schincaglia RM, Candow DG, Pimentel GD. Effect of Creatine Supplementation on Body Composition and Malnutrition-Inflammation Score in Hemodialysis Patients: An Exploratory 1-Year, Balanced, Double-Blind Design. Nutrients. 2024 Feb 23;16(5):615. doi: 10.3390/nu16050615. PMID 38474743
- [Background] Bossola M, Di Stasio E, Antocicco M, Pepe G, Tazza L, Zuccala G, Laudisio A. Functional impairment is associated with an increased risk of mortality in patients on chronic hemodialysis. BMC Nephrol. 2016 Jul 8;17(1):72. doi: 10.1186/s12882-016-0302-y. PMID 27391964
- [Background] Marini ACB, Pimentel GD. Is body weight or muscle strength correlated with the Malnutrition Inflammation Score (MIS)? A cross-sectional study in hemodialysis patients. Clin Nutr ESPEN. 2019 Oct;33:276-278. doi: 10.1016/j.clnesp.2019.07.009. Epub 2019 Aug 2. PMID 31451266
- [Background] Vanden Wyngaert K, Van Biesen W, Eloot S, Van Craenenbroeck AH, Calders P, Holvoet E. The importance of physical performance in the assessment of patients on haemodialysis: A survival analysis. PLoS One. 2022 May 19;17(5):e0268115. doi: 10.1371/journal.pone.0268115. eCollection 2022. PMID 35588129
- [Background] Daugirdas JT, Leypoldt JK, Akonur A, Greene T, Depner TA; FHN Trial Group. Improved equation for estimating single-pool Kt/V at higher dialysis frequencies. Nephrol Dial Transplant. 2013 Aug;28(8):2156-60. doi: 10.1093/ndt/gfs115. Epub 2012 May 4. PMID 22561585